CLINICAL TRIAL: NCT05541809
Title: Effect of Peppermint Aroma on Physiological Parameters of Mechanically Ventilated Patients
Brief Title: Peppermint Aroma and Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1532020
Record Dates: First submitted 2022-09-08; First posted 2022-09-15 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-09

CONDITIONS: Mechanical Ventilation Complication
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peppermint group (Experimental): This group will receive peppermint oil aroma
  Interventions: Other: Aromatherapy
- Water group (Placebo Comparator): This group will receive water as an aroma oil
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy — Peppermint aroma inhalation
  Arms: Peppermint group
Other: Placebo — Water inhalation
  Arms: Water group

SUMMARY:
Three drops of peppermint oil will be dropped on a cotton ball that will be fixed in the patient's collar. In the placebo group, peppermint oil will be replaced with water.

DETAILED DESCRIPTION:
Mechanical ventilathetion increases the anxiety of critically ill patients. The physiological parameters of those patients are affected by stress. Peppermint inhalation reduces stress and improves physiological parameters in many studies, but none of these studies used peppermint inhalation on mechanically ventilated patients.

Patients who are conscious on mechanical ventilation via endotracheal via tube will be randomly assigned to two groups. Patients will be kept intubated and mechanically ventilated. Nothing will be changed in patients' mechanical ventilation data. The intervention group will receive peppermint inhalation intervention, and the placebo group received water inhalation intervention. Patients in both groups will be assessed for their smell ability by Sniffin Sticks-test before starting the interventions.

Three drops of undiluted peppermint oil will be dropped on a cotton ball. Then it will be placed about 20 cm from the patient's nose. It will be fixed on the patient's collar. In the placebo group, the cotton ball will be soaked in water. Then, patients will be monitored for one hour.

ELIGIBILITY:
Inclusion Criteria: Patients with

* (1) endotracheal tube (ETT)
* (2) mechanical ventilation with spontaneous breathing modes which are CPAP, PIPAP and PSV
* (3) FOUR score equal to or more than 13,
* (4) RASS score from -1 to +4.

Exclusion Criteria: Patients with

* (1) respiratory asthma
* (2) chronic obstructive pulmonary disease
* (3) acute respiratory distress syndrome,
* Sniffin' Sticks-test score of smell less than 17

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | Change from baseline heart rate at one hour.
  The number of heart beats in one minute. It will be reported in beat per minute.
Respiratory rate | Change from baseline respiratory rate at one hour.
  The number of breaths in one minute. It will be reported in breath per minute.
Mean blood pressure | Change from baseline mean blood pressure at one hour.
  Mean blood pressure equal diastolic blood pressure + 1/3 [systolic blood pressure - diastolic blood pressure]. It will be reported in millimeters of mercury (mmHg).
Pain score | Change from baseline pain score at one hour.
  It will be measured using non verbal pain assessment scale. It consists of five categories; face, movement, guarding, physiology, and respiratory items. It will be reported in score. The maximum score of the scale is 10 which means extremely sever pain, and the minimum score is zero which means no pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Faculty of nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
No sharing of the patient data was planned